CLINICAL TRIAL: NCT01793584
Title: Randomized Trial of Laparoscopic Versus Abdominal Hysterectomy for Benign Indications and Impact on Surgical Success
Brief Title: Surgical Success After Laparoscopic vs Abdominal Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Kinberly Kho, Associate Professor, Department of Obstetrics and Gynecology, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STU 032012-067
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Metrorrhagia; Menorrhagia; Leiomyoma; Adenomyosis; Pelvic Pain; Endometriosis; Pelvic Inflammatory Disease
Keywords: Comparative effectiveness; Surgical success
MeSH Terms: conditions — Metrorrhagia; Menorrhagia; Leiomyoma; Adenomyosis; Pelvic Pain; Endometriosis; Pelvic Inflammatory Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopic hysterectomy (Active Comparator): Total laparoscopic hysterectomy, laparoscopic assisted vaginal hysterectomy
  Interventions: Procedure: Laparoscopic hysterectomy
- Abdominal hysterectomy (Active Comparator): Total Abdominal Hysterectomy
  Interventions: Procedure: Abdominal hysterectomy

INTERVENTIONS:
Procedure: Laparoscopic hysterectomy — LAVH, TLH
  Arms: Laparoscopic hysterectomy
Procedure: Abdominal hysterectomy — TAH
  Arms: Abdominal hysterectomy

SUMMARY:
The purpose of the proposed pilot study is to investigate the effectiveness, cost, safety, and long-term impact on quality of life of laparoscopic hysterectomy (LH) in relation to abdominal hysterectomy (AH) for the treatment of benign gynecologic disease in women through a randomized surgical trial.

DETAILED DESCRIPTION:
The overall hypothesis is that neither mode of hysterectomy will be consistently superior to the other with respect to each of the three domains of complications, cost, and patient-centered outcomes. The overall goal of the study is to determine which clinically relevant factors may impact the choice of LH compared to AH. The results of the study may be useful for clinicians, patients, hospital administrators and health policy makers.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing hysterectomy for benign indications within 8 weeks of enrollment
* Women >18 years of age
* Non-emergent surgery
* Non-pregnant

Exclusion Criteria:

* Candidate for vaginal hysterectomy
* Uterine size >14 weeks by clinical exam OR >300 mL by ultrasound measurement
* History of cancer of reproductive tract
* Requires concomitant pelvic organ prolapse (POP) surgery
* Requires surgery for urinary incontinence
* Has acute angle glaucoma
* Has severe cardiac/respiratory disease
* Desires supracervical hysterectomy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-02; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Quality of life | 1 year
  1) Patient-centered outcomes composite
  1. Quality of life - measured using the Short Form 12 (SF-12v2),
  2. Sexual functioning - measured using the Sexual Activity Questionnaire (SAQ)
  3. Body image - measured using the Body Image Scale (BIS)
  4. Return to normal activity -measured using the Activities Assessment Scale (AAS)
  5. Pain - measured using a 10 point likert scale
  6. Productivity - measured using a questionnaire about missed work

SECONDARY OUTCOMES:
Cost | 1 year
  Hospital charges and indirect costs of missed work/caregiving due to hysterectomy will be calculated
Complications | 1 year
  Intraoperative and postoperative complications including conversions, unintentional lacerations/injury to organs, hemorrhage, infection, wound complications, VTE, death, pain, neuropathy

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Kho, MD, MPH, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Hospital, Dallas, Texas, United States